CLINICAL TRIAL: NCT07022340
Title: Investigating Resistance Training for Vascular Function and Quality of Life in Perimenopausal Women
Brief Title: Hemodynamics After Resistance Training
Acronym: HeART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Marnie McLean, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00264586
Record Dates: First submitted 2025-06-04; First posted 2025-06-15 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Perimenopause
Keywords: menopause; perimenopause; vascular function; arterial stiffness; endothelial function; resistance exercise training; strength training; mood; sleep; quality of life; cardiovascular disease; estrogen deficiency; exercise
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance Training Intervention (Experimental): Participants randomized to resistance training will complete two sessions/week for 16 weeks.
  Interventions: Behavioral: Resistance Training Intervention
- Health Education Intervention (No Intervention): Participants randomized to the health education control group will receive weekly emails with general menopause information. They will be instructed to maintain current lifestyle habits, including exercise habits while enrolled in this study. They will be provided with a personalized resistance training program, equipment orientation/training session, and a counseling phone call with an exercise physiologist following study completion, or they can re-enroll in the resistance training intervention after completing the control portion of the study.

INTERVENTIONS:
Behavioral: Resistance Training Intervention — Participants will complete a brief aerobic warm-up and dynamic stretching prior to each strength training session. Participants will complete 9 exercises for all major muscle groups. Strength testing at the baseline study visit will be used to determine initial load. Participants will complete 1 set of moderate-intensity loads (~50% maximum and ~12 repetitions) in week 1, 2 sets in week 2, and 3 sets in week 3. By week 4, participants will be completing 3 sets at 60% of maximum. Weight loads will be progressively increased so volitional fatigue is reached by 8-12 repetitions/set.
  Arms: Resistance Training Intervention

SUMMARY:
Women's blood vessel health gets worse after menopause, or "the change of life". Some women exercise less during menopause. Exercise can improve blood vessel health. The investigators want to know if resistance exercise, like lifting weights, can improve blood vessel health in women who are just starting menopause. The investigators also want to know if lifting weights can improve mood, sleep, and quality of life in women going through menopause. The investigators will have two groups of women for this study. One group will lift weights (do resistance exercise) twice per week, and the other group will get emails with information about menopause. The investigators will measure blood vessel health, sleep, mood, and menopause symptoms at the start and the end of this study and compare women who did and did not exercise.

DETAILED DESCRIPTION:
Perimenopause is an important time when heart disease risk increases. Perimenopause is also related to worse health-related quality of life, sleep disruptions, and mood. Poor sleep and mood are both related to cardiovascular disease risk. Resistance exercise is effective at reducing cardiovascular disease risk in premenopausal women, and also improves mood, menopausal symptoms, and sleep quality in post-menopausal women. Resistance exercise does not consistently improve vascular function, such as arterial stiffness and blood vessel reactivity, in post-menopausal women. This study aims to investigate the effect of resistance training intervention on vascular function in perimenopausal women. This study will also determine if resistance training improves other novel cardiovascular disease risk factors that tend to worsen in perimenopause, such as sleep quality, mood, and menopause-specific quality of life.

The investigators will conduct a randomized controlled trial in perimenopausal females. Participants will complete baseline vascular function and exercise testing at baseline. Blood and urine will be collected. Participants will also complete surveys about their sleep, mood, and menopause-specific quality of life. Participants will be randomized to resistance training or control group. Those randomized to resistance training will complete two sessions per week for 16 weeks. The control group will receive a weekly health education email. Following the 16-week intervention or control, participants will complete post-intervention vascular function and exercise testing, and the same surveys as at baseline. Comparisons will be made between the exercise and control groups.

ELIGIBILITY:
* Are between 40-60 years old
* Have had menstrual irregularities in the last 12 months
* Do not currently complete more than two 30-min sessions of structured exercise per week and do not do any resistance training exercise;
* Are not currently pregnant
* Do not smoke or vape nicotine or marijuana
* Have not had an oophorectomy, hysterectomy, or surgical menopause
* Are not currently taking hormone replacement therapy
* Have not taken hormone replacement therapy in the last 6 months
* Are not taking steroidal medication or medication to treat diabetes, cholesterol, or high blood pressure
* Are able to exercise - your doctor has not told you that you cannot exercise
* Can attend a morning study visit at the University of Michigan's School of Kinesiology Building
* Are willing to avoid food 2 hours prior to the morning study visit
* Are willing to avoid strenuous exercise, caffeine, and alcohol, 8 hours prior to the morning study visit
* Are willing to participate in an exercise training program or health education program for 16 weeks

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Vascular function | At baseline and the end of the 16 week study period
  Arterial stiffness and wave reflection will be measured at baseline and following the 16-week study period using cuff-based waveform acquisition and applanation tonometry.
Endothelial Function | At baseline and the end of the 16 week study period
  Endothelial function will be measured at baseline and following the 16-week study period using brachial artery flow-mediated dilation measured with vascular ultrasound.

SECONDARY OUTCOMES:
Mood scores | At baseline and the end of the 16 week study period
  Mood will be assessed using validated surveys (PROMIS) at baseline and following the 16-week study period.
Sleep quality | At baseline and the end of the 16 week study period
  Sleep quality will be assessed using a validated survey (PSQI) at baseline and following the 16-week study period.
Menopause-specific quality of life | At baseline and the end of the 16 week study period
  Menopause-specific quality of life will be assessed using a validated survey (MENQOL) at baseline and following the 16-week study period

CONTACTS AND LOCATIONS:
Overall Officials: Marnie K. McLean, M.S., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Kinesiology, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Only deidentified data may be shared. No individual's name or identifiers will be published or shared. Requests for limited datasets will be considered.